CLINICAL TRIAL: NCT02890303
Title: A Prospective Multi-Center Study of Anterior Lens Capsulotomy Using the Mynosys Zepto System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mynosys Cellular Devices, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MYN-002
Record Dates: First submitted 2016-08-31; First posted 2016-09-07 (Estimated); Results first posted 2018-04-27 (Actual); Last update posted 2018-04-27 (Actual); Status verified 2018-04

CONDITIONS: Cataract
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Zepto Capsulotomy (Experimental): This study will evaluate outcome in subjects who have elected to have Zepto capsulotomies during cataract surgery. Effectiveness Rate - An effectiveness rate of 95% complete capsulotomies provides reasonable assurance that the Zepto system is effective. Primary Safety Endpoint - Posterior Capsular Rupture & Vitreous Loss (4% or less)
  Interventions: Device: Zepto System

INTERVENTIONS:
Device: Zepto System — Anterior Capsulotomy using the Zepto System.
  Other Names: Zepto

SUMMARY:
This study will evaluate outcome in subjects who have elected to have Zepto capsulotomies during cataract surgery with phacoemulsification.

DETAILED DESCRIPTION:
This study will evaluate outcome in subjects who have elected to have Zepto capsulotomies during cataract surgery with phacoemulsification to evaluate safety and effectiveness. The primary effectiveness endpoint is a complete capsulotomy in at least 95 percent of the cases. The primary safety endpoint is posterior capsular rupture and virtuous loss in 4 percent or less of the subjects. Other parameters to be captured during the study include anterior capsule tears, corneal touch, capsulotomy diameter, contraption of the Zepto capsulotomy, size of the corneal incision pre and post Zepto, interocular lens contraption and evaluation of zonular stability and the incidence and severity of adverse events. The criteria for patient success will be accessed based on the successful completion of a 360 degree capsulotomy without tissue bridges and no posterior capsule rupture and vitreous loss. The criteria for study success will be accessed based on a greater than or equal to 95 percent of the cases having a complete 360 degree capsulotomy without tissue bridges and less than 4 percent of subjects with posterior capsule rupture and vitreous loss.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must be age 22 or older,
2. Subjects consenting to undergoing phacoemulsification and IOL implant surgery for the treatment of symptomatic age related lens cataract, and then electing to undergo ZeptoTM capsulotomy,
3. Subjects must be willing and able to return for scheduled treatment and follow-up examinations for 3 months.

Exclusion Criteria:

1. Disease or pathology in the treatment eye that will compromise visual performance or refractive outcome (e.g. previous refractive surgery),
2. Zonular abnormality,
3. Posterior polar cataract,
4. Fellow eye with acuity less than 20/200,
5. Any prior ocular surgery of the study eye,
6. Pupillary dilation during the pre-operative exam of less than 7 mm in diameter,
7. Proliferative diabetic retinopathy,
8. Disorders of the ocular muscles, such as nystagmus or strabismus,
9. Chronic uveitis,
10. Abnormal corneal endothelium,
11. Subjects on medications with, in the opinion of the surgeon, significant ocular side effects,
12. Pregnant or nursing (lactating) women,
13. Implanted ocular device or drug in the study eye,
14. Any other condition, which in the judgment of the investigator would prevent the subject from completing the study (e.g. documented diagnosis or treatment for symptoms associated with dementia, mental illness),
15. Current participation in another drug or device clinical study, or participation in such a clinical study within the six months.

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2016-09-12 (Actual); Primary Completion 2016-12-15 (Actual); Study Completion 2017-03-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William Christie, M.D., Principal Investigator — Scott & Christie and Associates P C; Daniel H Chang, M.D., Principal Investigator — Empire Eye and Laser Center; David F Chang, M.D., Principal Investigator — Peninsula Eye Surgery Center; Eric D Donnenfeld, M.D., Principal Investigator — Lasik Garden City; Philip C Hoopes, M.D., Principal Investigator — Hoopes Vision; John Vukich, M.D., Principal Investigator — Davis Duehr Dean Clinic; Farrell C Tyson II, M.D., Principal Investigator — Cape Coral Eye Ctr Pa; Vance Thompson, M.D, Principal Investigator — Vance Thompson Vision

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chang DF, Mamalis N, Werner L. Precision Pulse Capsulotomy: Preclinical Safety and Performance of a New Capsulotomy Technology. Ophthalmology. 2016 Feb;123(2):255-264. doi: 10.1016/j.ophtha.2015.10.008. Epub 2015 Nov 12. PMID 26578447
- [Background] Carifi G, Miller MH, Pitsas C, Zygoura V, Deshmukh RR, Kopsachilis N, Maurino V. Complications and outcomes of phacoemulsification cataract surgery complicated by anterior capsule tear. Am J Ophthalmol. 2015 Mar;159(3):463-9. doi: 10.1016/j.ajo.2014.11.027. Epub 2014 Nov 26. PMID 25461300
- [Background] Agrawal V, Upadhyay J; Indian Cataract Risk Stratification Study group. Validation of scoring system for preoperative stratification of intra-operative risks of complications during cataract surgery: Indian multi-centric study. Indian J Ophthalmol. 2009 May-Jun;57(3):213-5. doi: 10.4103/0301-4738.49396. PMID 19384016
- [Background] Ang GS, Whyte IF. Effect and outcomes of posterior capsule rupture in a district general hospital setting. J Cataract Refract Surg. 2006 Apr;32(4):623-7. doi: 10.1016/j.jcrs.2006.01.047. PMID 16698484
- [Background] Chan FM, Mathur R, Ku JJ, Chen C, Chan SP, Yong VS, Au Eong KG. Short-term outcomes in eyes with posterior capsule rupture during cataract surgery. J Cataract Refract Surg. 2003 Mar;29(3):537-41. doi: 10.1016/s0886-3350(02)01622-x. PMID 12663021
- [Background] Desai P, Minassian DC, Reidy A. National cataract surgery survey 1997-8: a report of the results of the clinical outcomes. Br J Ophthalmol. 1999 Dec;83(12):1336-40. doi: 10.1136/bjo.83.12.1336. PMID 10574810
- [Background] Greenberg PB, Tseng VL, Wu WC, Liu J, Jiang L, Chen CK, Scott IU, Friedmann PD. Prevalence and predictors of ocular complications associated with cataract surgery in United States veterans. Ophthalmology. 2011 Mar;118(3):507-14. doi: 10.1016/j.ophtha.2010.07.023. Epub 2010 Oct 29. PMID 21035868
- [Background] Hyams M, Mathalone N, Herskovitz M, Hod Y, Israeli D, Geyer O. Intraoperative complications of phacoemulsification in eyes with and without pseudoexfoliation. J Cataract Refract Surg. 2005 May;31(5):1002-5. doi: 10.1016/j.jcrs.2004.09.051. PMID 15975469
- [Background] Ionides A, Minassian D, Tuft S. Visual outcome following posterior capsule rupture during cataract surgery. Br J Ophthalmol. 2001 Feb;85(2):222-4. doi: 10.1136/bjo.85.2.222. PMID 11159491
- [Background] Lundstrom M, Barry P, Leite E, Seward H, Stenevi U. 1998 European Cataract Outcome Study: report from the European Cataract Outcome Study Group. J Cataract Refract Surg. 2001 Aug;27(8):1176-84. doi: 10.1016/s0886-3350(01)00772-6. PMID 11524187
- [Background] Martin KR, Burton RL. The phacoemulsification learning curve: per-operative complications in the first 3000 cases of an experienced surgeon. Eye (Lond). 2000 Apr;14 ( Pt 2):190-5. doi: 10.1038/eye.2000.52. PMID 10845015
- [Background] Zaidi FH, Corbett MC, Burton BJ, Bloom PA. Raising the benchmark for the 21st century--the 1000 cataract operations audit and survey: outcomes, consultant-supervised training and sourcing NHS choice. Br J Ophthalmol. 2007 Jun;91(6):731-6. doi: 10.1136/bjo.2006.104216. Epub 2006 Oct 18. PMID 17050577
- [Background] Simanovskii DM, Mackanos MA, Irani AR, O'Connell-Rodwell CE, Contag CH, Schwettman HA, Palanker DV. Cellular tolerance to pulsed hyperthermia. Phys Rev E Stat Nonlin Soft Matter Phys. 2006 Jul;74(1 Pt 1):011915. doi: 10.1103/PhysRevE.74.011915. Epub 2006 Jul 24. PMID 16907135
- [Background] Thompson VM, Berdahl JP, Solano JM, Chang DF. Comparison of Manual, Femtosecond Laser, and Precision Pulse Capsulotomy Edge Tear Strength in Paired Human Cadaver Eyes. Ophthalmology. 2016 Feb;123(2):265-274. doi: 10.1016/j.ophtha.2015.10.019. Epub 2015 Dec 23. PMID 26707416
- [Background] Auffarth GU, Reddy KP, Ritter R, Holzer MP, Rabsilber TM. Comparison of the maximum applicable stretch force after femtosecond laser-assisted and manual anterior capsulotomy. J Cataract Refract Surg. 2013 Jan;39(1):105-109. doi: 10.1016/j.jcrs.2012.08.065. PMID 23245363
- [Background] Nagy Z, Takacs A, Filkorn T, Sarayba M. Initial clinical evaluation of an intraocular femtosecond laser in cataract surgery. J Refract Surg. 2009 Dec;25(12):1053-60. doi: 10.3928/1081597X-20091117-04. PMID 20000286
- [Background] Trivedi RH, Wilson ME Jr, Bartholomew LR. Extensibility and scanning electron microscopy evaluation of 5 pediatric anterior capsulotomy techniques in a porcine model. J Cataract Refract Surg. 2006 Jul;32(7):1206-13. doi: 10.1016/j.jcrs.2005.12.144. PMID 16857511
- [Background] Androudi S, Brazitikos PD, Papadopoulos NT, Dereklis D, Symeon L, Stangos N. Posterior capsule rupture and vitreous loss during phacoemulsification with or without the use of an anterior chamber maintainer. J Cataract Refract Surg. 2004 Feb;30(2):449-52. doi: 10.1016/S0886-3350(03)00584-4. PMID 15030840
- [Background] Mearza AA, Ramanathan S, Bidgood P, Horgan S. Visual outcome in cataract surgery complicated by vitreous loss in a district general hospital. Int Ophthalmol. 2009 Jun;29(3):157-60. doi: 10.1007/s10792-008-9214-6. Epub 2008 Apr 10. PMID 18401555
- [Background] Tan JH, Karwatowski WS. Phacoemulsification cataract surgery and unplanned anterior vitrectomy--is it bad news? Eye (Lond). 2002 Mar;16(2):117-20. doi: 10.1038/sj.eye.6700015. PMID 11988808
- [Background] Chang JS, Chen IN, Chan WM, Ng JC, Chan VK, Law AK. Initial evaluation of a femtosecond laser system in cataract surgery. J Cataract Refract Surg. 2014 Jan;40(1):29-36. doi: 10.1016/j.jcrs.2013.08.045. Epub 2013 Nov 22. PMID 24269139
- [Background] Nagy ZZ, Takacs AI, Filkorn T, Kranitz K, Gyenes A, Juhasz E, Sandor GL, Kovacs I, Juhasz T, Slade S. Complications of femtosecond laser-assisted cataract surgery. J Cataract Refract Surg. 2014 Jan;40(1):20-8. doi: 10.1016/j.jcrs.2013.08.046. PMID 24355719
- [Background] Roberts TV, Lawless M, Bali SJ, Hodge C, Sutton G. Surgical outcomes and safety of femtosecond laser cataract surgery: a prospective study of 1500 consecutive cases. Ophthalmology. 2013 Feb;120(2):227-33. doi: 10.1016/j.ophtha.2012.10.026. Epub 2012 Dec 6. PMID 23218822

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study enrolled patients at 8 clinical study sites, with symptomatic age-related lens cataract desiring lens extraction and IOL implantation. The last patient was enrolled in the study in December 2016.
Period: Overall Study
Arm/Group | Zepto Capsulotomy
Started | 100
Completed | 100
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Zepto Capsulotomy
Number analyzed (Participants) | 100
Age, Customized [Mean (Full Range); unit: years] | 69.4 [46 to 89]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 58
  Male | 42
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 92
  More than one race | 0
  Unknown or Not Reported | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 100
Intraocular Pressure [Mean (Full Range); unit: mm Hg] | 16 [7 to 35]
Manifest Refraction [Count of Participants; unit: Participants] | 96
Uncorrected distance visual acuity (UCVA) [Mean (Full Range); unit: ft] | 138 [25 to 800]
Best spectacle corrected distance visual acuity (BSCVA) [Mean (Full Range); unit: ft] | 40 [20 to 400]
Slit Lamp [Number; unit: percentage of participants]
  % of Normal treatment lids | 97
  % presenting with 1 + Meibomian gland dysfunction | 7
  % of Normal cornea | 97
  % 1 + punctuate epithelial keratitis/ keratopathy | 1
  % with Waite Beecham Lines - mild | 1
  % with faint stromal scarring | 1
Fundus Examination [Number; unit: percentage of participants]
  % with normal findings | 87
  % presented with posterior vitreous detachment | 7
  % with mild macular drusen | 1
  % with peripheral drusen | 1
  % with mild epiretinal membrane | 1
  % with choroidal nevus | 1
  % with post vitreous degeneration | 1
  % with a tilted disc | 1
Dilated Pupil Size [Mean (Full Range); unit: mm] | 8 [6 to 9.5]

OUTCOME MEASURES:

1. Primary Outcome: Complete Capsulotomy
Description: A successful complete Zepto capsulotomy is defined in this protocol to be one that results in a complete 360 degree capsulotomy without any residual tissue bridges visible to the surgeon. If there are such tissue bridges, the surgeon completes the capsulotomy manually.
  The primary effectiveness endpoint was defined as :Complete capsulotomy (target ≥ 95% of cases).
Time Frame: During surgery
Measure: Number; unit: participants
Arm/Group | Zepto Capsulotomy
Number analyzed (Participants) | 100
participants | 98

ADVERSE EVENTS:
Time Frame: Adverse event data will be collected from Day 0 (once the Informed Consent Form has been signed) until 1 month post surgery. Data points include Day 0, Day 1, 1 week and 1 month post-op.
Arm/Group | Zepto Capsulotomy
All-Cause Mortality (participants affected / at risk) | 0/100
Serious Adverse Events (participants affected / at risk) | 0/100
Other Adverse Events (participants affected / at risk) | 5/100
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Zepto Capsulotomy (N=100)
Epithelial Erosion (Eye disorders) | 1 (1)
Macular Edema (Eye disorders) | 1 (1)
Anterior Capsule Tear (Eye disorders) | 2 (2)
Posterior Tear without Vitreous Loss (Eye disorders) | 1 (1)
Headache (General disorders) | 1 (1)
Elevated IOP (Eye disorders) | 1 (1)
Ache in Treatment Eye (Eye disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2016-07-06): https://cdn.clinicaltrials.gov/large-docs/03/NCT02890303/Prot_000.pdf
  • Informed Consent Form (2016-09-08): https://cdn.clinicaltrials.gov/large-docs/03/NCT02890303/ICF_001.pdf